CLINICAL TRIAL: NCT05441488
Title: A 96-Week, Prospective, Multicenter, Randomised, Double-Blind, Placebo-Controlled, Phase 3 Study to Compare Efficacy and Safety of Masitinib Dose Titration to 4.5 mg/kg/Day Versus Placebo in the Treatment of Patients With Primary Progressive or Secondary Progressive Multiple Sclerosis Without Relapse
Brief Title: Masitinib in the Treatment of Patients With Primary Progressive or Non-active Secondary Progressive Multiple Sclerosis
Acronym: MAXIMS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB20009; MAXIMS
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Primary progressive MS; Non-active secondary progressive MS; Tyrosine kinase inhibitor; PPMS; SPMS
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Masitinib (4.5) (Experimental): Participants receive masitinib (3.0 mg/kg/day), given orally twice daily, with a dose escalation to 4.5 mg/kg/day after 4 weeks of treatment. Each ascending dose titration is subjected to a safety control.
  Interventions: Drug: Masitinib (4.5)
- Placebo (Placebo Comparator): Participants receive a matched dose placebo, given orally twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — treatment per os
  Other Names: Placebo Oral Tablet
  Arms: Placebo
Drug: Masitinib (4.5) — Masitinib (titration to 4.5 mg/kg/day)
  Other Names: AB1010
  Arms: Masitinib (4.5)

SUMMARY:
To evaluate the efficacy and safety of oral masitinib versus placebo in the treatment of patients with primary progressive or secondary progressive multiple sclerosis without relapse.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor, targeting innate immune cells (mast cells and microglia) that are involved in the pathophysiology of progressive multiple sclerosis (MS). This is a multicenter, double-blind, randomized, placebo-controlled, comparative study of oral masitinib in the treatment of patients with progressive MS who were progressing but not clinically active.

ELIGIBILITY:
Main inclusion criteria include:

* Patients with either primary progressive or secondary progressive multiple sclerosis with onset of symptoms at least five years before baseline and with no relapse diagnosed according to the 2017 revised McDonald's criteria at least two years before screening
* Patients with Expanded Disability Status Scale (EDSS) score between 3.0 to 6.0 (both inclusive) at screening and baseline
* Patients with an EDSS score progression ≥1 point with no improvement during 2 years
* Absence of T1 Gadolinium-enhancing brain lesions as measured by MRI at screening

Main exclusion criteria include:

* Patients suffering from a disease other than MS that would better explain the patient's neurological clinical signs and symptoms and/or MRI lesions observed at screening
* Inability to complete screening MRI (contraindications for MRI) and/or any known allergy or hypersensitivity or any contra-indication to gadolinium macrocyclic
* Patients treated with other disease modifying treatments in the time frames and conditions mentioned under previous treatment wash out period, assessed at baseline
* Patients with lymphocytes <1.0 × 10^9/L at screening and at baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Time to confirmed progression | 96 weeks
  Time to disability progression, confirmed by two consecutive visits, wherein progression of disability is measured by the Expanded Disability Status Scale (EDSS) with progression defined as a 1-point worsening for baseline EDSS score ≤5.5, or 0.5-point worsening for baseline EDSS score >5.5.
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The EDSS provides a total score on a scale that ranges from 0 to 10, in 0.5-point increments, with higher scores indicating greater disability. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.

SECONDARY OUTCOMES:
Time to Expanded Disability Status Scale (EDSS) score of 7.0 | 96 weeks
  Time to reach EDSS score of 7 from baseline up to week 96, wherein EDSS score of ≥7.0 represents wheelchair dependency.
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The EDSS provides a total score on a scale that ranges from 0 to 10, in 0.5-point increments, with higher scores indicating greater disability. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.
Overall Change in Expanded Disability Status Scale (EDSS) Score | 96 weeks
  Change from baseline on the EDSS, calculated using repeated measures methodology on all time points measured over 96 weeks (i.e., a population-averaged score comprising consecutive data points from each patient).
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The EDSS provides a total score on a scale that ranges from 0 to 10, in 0.5-point increments, with higher scores indicating greater disability. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.
Brain Magnetic Resonance Imaging Assessments | 96 weeks
  Change in baseline brain volume and lesions will be measured and assessed
Multiple Sclerosis Quality of Life (MSQOL)-54 | 96 weeks
  Change in quality of life assessment instrument MSQOL-54 The MS Quality of Life Instrument (MSQoL-54) is a structured self-report questionnaire that is used to assess the impact of MS on the individual's well-being. It consists of 52 items combined in 12 subscales, and two single items. Higher scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick VERMERSCH, MD, PhD, Principal Investigator — University of Lille, CHU of Lille, France
Locations (37):
- France (9):
  - Service de Neurologie Hôpital Henri-Mondor, Créteil
  - Hôpital Roger Salengro, Lille
  - Hôpital Pasteur - CHU de Nice, Nice
  - Centre Hospitalier Universitaire Nimes - Service de Neurologie, Nîmes
  - Centre hospitalier intercommunal de Poissy-Saint-Germain-en-Laye, Poissy
  - Le Centre hospitalier universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Centre Hospitalier Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire Toulouse, Toulouse
- Greece (5):
  - Athens Naval Hospital, Athens
  - Eginition Hospital, Athens University Medical School, Athens
  - General University Hospital of Larissa, Larissa
  - AHEPA University Hospital, Aristotle University of Thessaloniki, Thessaloniki
  - Private Clinic ELPIS, Volos
- Azienda Ospedaliero Universitaria Policlinico "G.Rodolico -San Marco", Catania, Italy
- Poland (7):
  - Nzoz Neuro-Medic, Katowice
  - NOVI-MED, Ksawerów
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - NZOZ Neuro-Med, Lublin
  - Generała Jarosława Dąbrowskiego, Oświęcim
  - NZOZ Neuro-Kard, Poznan
  - Clinical Best Solutions, Warsaw
- Russia (4):
  - State Budgetary Institution of Health of the City of Moscow City Polyclinic #2, Moscow
  - Perm Regional Clinical Hospital, Perm
  - City Hospital No. 40 Kurortny District, Saint Petersburg
  - LLC "Center of socially significant diseases", Saint Petersburg
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Gregorio Marañón General University Hospital, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Centrum för neurologi, Stockholm
- Ukraine (4):
  - Lviv Regional Clinical Hospital, Lviv
  - Rivne Regional Specialized Dispensary for Radiation Protection of the Population Municipal Enterprise, Rivne
  - Communal Non-Profit Enterprise "Ternopil Regional Clinical Psychoneurological Hospital" of Ternopil Regional Council, Department of Neurology #1, Ternopil
  - Salutem Medical Center, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vermersch P, Brieva-Ruiz L, Fox RJ, Paul F, Ramio-Torrenta L, Schwab M, Moussy A, Mansfield C, Hermine O, Maciejowski M; AB07002 Study Group. Efficacy and Safety of Masitinib in Progressive Forms of Multiple Sclerosis: A Randomized, Phase 3, Clinical Trial. Neurol Neuroimmunol Neuroinflamm. 2022 Feb 21;9(3):e1148. doi: 10.1212/NXI.0000000000001148. Print 2022 May. PMID 35190477
- [Background] Vermersch P, Benrabah R, Schmidt N, Zephir H, Clavelou P, Vongsouthi C, Dubreuil P, Moussy A, Hermine O. Masitinib treatment in patients with progressive multiple sclerosis: a randomized pilot study. BMC Neurol. 2012 Jun 12;12:36. doi: 10.1186/1471-2377-12-36. PMID 22691628
- [Derived] Latham BD, Oskin DS, Crouch RD, Vergne MJ, Jackson KD. Cytochromes P450 2C8 and 3A Catalyze the Metabolic Activation of the Tyrosine Kinase Inhibitor Masitinib. Chem Res Toxicol. 2022 Sep 19;35(9):1467-1481. doi: 10.1021/acs.chemrestox.2c00057. Epub 2022 Sep 1. PMID 36048877